CLINICAL TRIAL: NCT02216630
Title: An Open-label, Non-Randomized, Multi-center Study to Assess the Safety and Effects of Intravenous Implantation of Liposuction Derived Autologous Adipose-derived Stem Cells in Subjects With Chronic Obstructive Pulmonary Disease (COPD)
Brief Title: Safety and Efficacy of Adipose Derived Stem Cells for Chronic Obstructive Pulmonary Disease
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Kimera Society Inc (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: KS-SVF-1002
Record Dates: First submitted 2014-08-07; First posted 2014-08-15 (Estimated); Last update posted 2017-07-25 (Actual); Status verified 2017-07

CONDITIONS: Chronic Obstructive Pulmonary Disease
Keywords: COPD
MeSH Terms: conditions — Pulmonary Disease, Chronic Obstructive | interventions — Therapeutics

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Adipose-Derived Stem Cell (ADSC) Therapy (Experimental): This arm, as the sole arm, will consist of the ADSC treatment procedure. Intervention will consist of Adipose Derived Stem Cell (ADSC) Therapy
  Interventions: Drug: Adipose Derived Stem Cell (ADSC) Therapy

INTERVENTIONS:
Drug: Adipose Derived Stem Cell (ADSC) Therapy — Patients undergo a liposuction where 100 cc of fat are extracted. The ADSCs are then isolated and injected intravenously.

SUMMARY:
This will be an open-label, non-randomized multi-center study designed to assess the safety and efficacy of Adipose-derived Stem Cell (ASC) IV implantation. The therapy is composed of cells isolated from a patient's own adipose tissue. Liposuction will be performed to collect the adipose tissue specimen for subsequent processing to isolate the stem cells.

DETAILED DESCRIPTION:
In the context of the proposed study, adipose derived stem cells (ASC) constitute an autologous cell product that is delivered to the patient via intra-venous injection. In this study, we propose to investigate the immunosuppressive potential of the non-manipulated non-cultured stromal vascular fraction obtained via liposuction. Endpoints will be measured both by improvement of the forced evacuation volume in one second (FEV1) and distance covered in a 6 minute walk distance test (6MWD). The stromal vascular fraction comprises stromal cells isolated from total fat via enzymatic digestion ex-vivo. These cells are not cultured but are isolated from adipose tissue using a sterile tissue process in under two hours. The process includes rinsing in a saline solution to remove red blood cells, draining, and enzymatic digestion (collagenase) which isolates endothelial cells from adipose tissue. Post-processing, the pellet obtained via centrifugation is filtered and delivered to the patient who remains sedated within the same ambulatory center.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 to 85, inclusive
* A prior diagnosis of moderate to severe COPD
* GOLD IIa, III, IV

Exclusion Criteria:

* Pregnant or lactating
* Life expectancy < 6 months due to concomitant illnesses.
* Exposure to any investigational drug or procedure within 1 month prior to study entry or enrolled in a concurrent study that may confound results of this study.
* Any illness which, in the Investigators judgment, will interfere with the patient's ability to comply with the protocol, compromise patient safety, or interfere with the interpretation of study results
* Subjects on chronic immunosuppressive or chemotherapeutic therapy
* Known drug or alcohol dependence or any other factors which will interfere with the study conduct or interpretation of the results or who in the opinion of the investigator are not suitable to participate.
* Subjects with Alpha-1 antitrypsin deficiency (an inherited disorder that can cause lung disease and liver disease).
* Unwilling and/or not able to give written consent
* Patient is positive for hepatitis (past history of Hepatitis A is allowed)
* Any medical condition, which in the opinion of the clinical investigator, would interfere with the treatment or outcome of the patient
* Cerebral aneurysm clips

Ages: 18 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2014-08; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

PRIMARY OUTCOMES:
FEV1 Decline | 12 months
  The primary efficacy outcome will be a FEV1 decline of approximately or less than 30 ml at 12 month follow-up.
Number of Adverse Events | 12 months

SECONDARY OUTCOMES:
Secondary Efficacy Objective | 12 Months
  The secondary efficacy objective will be a decrease in six minute walking distance (6MWD) of less than 5% over one year.

CONTACTS AND LOCATIONS:
Locations (5):
- United States (5):
  - Melvin Propis M.D., Davie, Florida
  - Chicago, Chicago, Illinois
  - Las Vegas, Las Vegas, Nevada
  - New York, New York, New York
  - Dallas, Dallas, Texas